CLINICAL TRIAL: NCT01895751
Title: A Clinical Trial of Conservative Versus Routine Invasive Management in Patients with Prior Coronary Artery Bypass Surgery in Patients with a Non-ST Elevation Acute Coronary Syndrome: a Pilot Trial and Registry.
Brief Title: Conservative Non-Invasive Versus Routine Invasive Management in Coronary Artery Bypass Surgery Patients with Non ST Elevation Elevation Acute Coronary Syndrome
Acronym: CABG-ACS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NHS National Waiting Times Centre Board (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Principal Investigator, Colin Berry, Professor Colin Berry, NHS National Waiting Times Centre Board
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GN-11-CA456
Record Dates: First submitted 2013-05-24; First posted 2013-07-10 (Estimated); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Non ST Elevation Myocardial Infarction; Unstable Angina
Keywords: Non-ST elevation myocardial infarction (NSTEMI); Non-ST elevation acute coronary syndrome (NSTE-ACS); Unstable Angina; Medical therapy; Coronary angiogram; Percutaneous coronary intervention; Coronary artery bypass surgery; Coronary revascularization; Health economics
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction; Angina, Unstable

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conservative therapy (No Intervention): Conservative therapy group involves optimal medical therapy according to local hospital protocols with selective invasive management as clinically appropriate. Patients assigned to the conservative group may be referred for invasive management if the patient meets one of the following pre-specified criteria:
  Recurrent or refractory (class III or IV) angina with documented ischaemic ECG changes while on "optimal" medical therapy.
  New ST segment elevation in two contiguous leads without Q waves or T wave inversion greater than 3 mm or development of hemodynamic instability Deterioration in heart failure status (defined as Killip class 3 or 4).
- Invasive management (Active Comparator): Invasive management is timed as appropriate according to local NHS protocols. Usually, invasive management is expected to be performed in line with contemporary guidelines.
  Interventions: Procedure: Invasive management

INTERVENTIONS:
Procedure: Invasive management — Invasive management includes coronary and graft angiography (diagnostic imaging test) and coronary and/or graft revascularization with percutaneous coronary intervention (PCI) and/or coronary artery bypass graft (CABG), as clinically appropriate.
  Arms: Invasive management

SUMMARY:
Background: Most coronary artery bypass grafts (CABG) are diseased or blocked within 10 years of surgery meaning CABG survivors have an ever increasing risk of recurrent angina, heart attack and death. Given the large number of CABG survivors in the United Kingdom (UK), and the complexities of their clinical management, their heart health problems and related treatment are an increasing challenge in the UK National Health Service (NHS) and worldwide.

There is considerable controversy in the NHS and internationally about how to best manage patients with prior CABG and unstable angina / non-ST elevation acute coronary syndromes (NSTE-ACS). This is because there is no robust evidence to inform treatment practices or clinical guidelines since, historically, these patients have been excluded from randomised trials. This is the rationale for our study.

Aims: Our overall aim is to undertake a clinical trial of conservative non-invasive management with optimal drug therapy versus routine invasive management in NSTE-ACS patients with prior CABG during routine clinical care in NHS hospitals across the UK. Our trial is a proof-of-concept study of feasibility, safety, potential efficacy and health economics.

Hypothesis: A routine invasive approach in NSTE-ACS patients with prior CABG will not be superior to a conservative non-invasive approach with optimal medical therapy.

Design: The pilot study will involve 60 patients recruited in large urban hospitals (Western Infirmary, Glasgow Royal Infirmary) and district general hospitals (Royal Alexandra Hospital, Royal Blackburn Hospital (RBH)) to reflect usual practice in the UK. One of these hospitals (RBH) has an on-site cardiac catheterization laboratory, whereas the other hospitals refer patients who have been triaged for invasive management to the regional cardiothoracic centre (the Golden Jubilee National Hospital). In this proof of concept study, the investigators aim to gather information about screening, recruitment, randomisation, patient characteristics (including comorbidity and quality of life) and initial clinical outcomes to inform the design of the definitive trial. The follow-up will be in line with standard clinical care i.e. 30-42 days and 1 year. The investigators will hold data in the longer term to enable long-term follow-up analyses. The investigators will record information on NSTE-ACS patients with prior CABG who are ineligible to take part or who do not wish to be randomised as part of all follow-up registry of 'all-comers'.

DETAILED DESCRIPTION:
Background: Coronary artery bypass graft (CABG) surgery is commonly performed in the NHS and worldwide based on historical evidence of benefit over medical therapy and more recent evidence of benefit over percutaneous coronary intervention (PCI). According to the national audit data from the Society of Cardiothoracic Surgeons and the British Cardiovascular Intervention Society, over 1 million CABG operations have been performed in the UK, with 20,000 - 25,000 operations performed annually since 1994. Although the number of isolated CABG operations performed annually has fallen slightly (e.g. 17,822 in 2010), CABG combined with valve surgery has increased. Since the 5 year survival rate after CABG is approximately 90%, several hundred thousand patients with prior CABG are likely alive in the UK. However, occlusive vein graft disease affects around 10% of patients within 12 months of surgery and affects at least two thirds of patients by 10 years. Furthermore, disease in the native coronary arteries may also deteriorate. Consequently, even though vein graft occlusion may initially be subclinical, angina eventually recurs in most patients with repeat revascularisation (almost always by PCI) required in nearly two thirds of patients by 12 years. Furthermore, when PCI is performed in these patients clinical outcomes in the longer term are poor because of restenosis.

Given the large number of CABG survivors in the UK, and the complexities of their clinical management, their cardiac morbidity and mortality is an increasing challenge in NHS hospitals.

Chest pain is the commonest reason for hospital admission in the UK and more than 1 in 10 hospital admissions with suspected acute myocardial infarction (MI) have a history of prior CABG and non-ST elevation acute coronary syndrome (NSTE-ACS) patients with prior CABG spend more time in hospital than those without a history of CABG. According to the Myocardial Ischaemia National Audit Project (MINAP), 47,162 patients were admitted with an NSTE-ACS in England and Wales during 2009/2010 including approximately 5000 patients with prior CABG. The median 30-day death rate of all NSTE-ACS patients in the UK in 2009/2010 was approximately 7.5% and clinical outcomes in CABG patients are much worse than in patients without prior CABG. However, since prior CABG status is not an independent predictor of mortality, the prognostic determinants are multifactorial and strongly influenced by age and co-morbidity.

There is an important lack of evidence to inform clinical decision making in symptomatic CABG patients hospitalised with NSTE-ACS. Firstly, most clinical trials of treatment strategies in ACS have excluded patients with prior CABG. The pivotal clinical trials which specifically compared invasive versus conservative management in unstable coronary syndromes, including Thrombolysis in Myocardial Infarction (TIMI) IIIb, Fragmin during Instability in Coronary Artery Disease (FRISC) II, Treat Angina With Aggrastat and Determine the Cost of Therapy With an Invasive or Conservative Strategy (TACTICS)-TIMI 18, and Randomized Intervention Treatment of Angina (RITA) 3, excluded patients with prior CABG, meaning evidence is lacking on which treatment strategy is most appropriate in this patient group. In the absence of trial data, guidelines for clinicians are based on observational studies, a subgroup analysis and expert opinion (level of evidence C). According to the UK National Institute of Clinical Excellence (NICE) Clinical Guideline 94, "in the absence of more research, consensus expert opinion is the best that can be achieved." Although CABG patients with acute ischaemia are often managed invasively, angiography commonly does not lead to revascularisation. PCI, or even repeat CABG, is technically challenging, complications are common and longer term outcomes are poor. This is especially the case for repeat PCI in vein grafts. Overall, invasive management of patients with prior CABG is technically challenging and health outcomes are influenced by the effectiveness of the procedure and complications (safety). Procedural success is harder to achieve because of advanced native coronary and graft disease and co-morbidity meaning the procedure is less often a success and the risks of complications and adverse events (e.g. stroke) are three-four fold higher than average. Since the internal mammary graft is almost always patent, redo surgery is rarely performed because sternotomy may damage the mammary graft (which can be a life-threatening complication) and current guidelines recommend PCI unless the mammary graft is occluded.

The effectiveness of a routine invasive approach in every-day clinical practice, which is the approach of many clinicians, is called into question because acute and long term outcomes are much worse than in patients without prior CABG. PCI in redo CABG carries a four-fold higher risk of death compared to the index procedure and complications associated with PCI include bleeding, stroke and contrast nephropathy. Redo CABG confers a much higher risk than percutaneous coronary intervention (PCI). Overall, increased age and co-morbidity are common and key drivers of long-term outcome. Outcomes after PCI in vein grafts or native vessel disease are poor. For example, in Wales, of 161 patients who had PCI after CABG, adverse cardiac events occurred in 14% of them by 13 months (mainly related to repeat PCI (12%). In the UK overall, of 33,652 PCIs performed in 1999/2000, 907 (2.7%) were performed in patients with prior CABG. Only 1 in 10 procedures were reported as successful and 1.3% and 1.0% of patients experienced in-hospital MI or death. Ten years on (2009/2010), 8.4% of all patients undergoing PCI had a history of prior CABG and procedure-related outcomes remained disappointingly similar (1 in 10 procedures unsuccessful, in-hospital death rate (1.0%), 30-day mortality 1.5%).

By contrast, the efficacy of contemporary optimal medical therapies in patients with prior CABG is at least as good as in patients without prior CABG. Furthermore, medical therapy is not associated with procedure-related complications and potentially may be safer than invasive management. In contrast to revascularisation trials, patients with prior CABG are usually not excluded from contemporary drug trials (e.g. PLATO) and the evidence for secondary prevention medical therapies in patients with prior CABG is reasonably robust. In fact, some therapeutic trials have specifically focused on post-CABG patients and have shown that statin therapy attenuates graft disease progression and improves patient outcomes. In ACS patients with prior CABG, health outcomes are also improved by treatment with contemporary anti-platelet drug therapies. New evidence-based medicines continue to emerge including more potent anti-platelet drugs such as ticagrelor and prasugrel and safer anti-coagulants, such as fondaparinux. Our strategy is also predicated on use of optimal anti-ischaemic therapies, including novel drugs such as ivabradine, as clinically appropriate.

PRACTICES AND UNCERTAINITIES ASSOCIATED WITH MANAGEMENT OF CABG PATIENTS WITH ACUTE ISCHEMIA: Since most patients with prior CABG and an acute NSTE-ACS will be intermediate-high risk, most patients will be considered for invasive management according to guideline recommendations. Registries indicate that invasive management only occurs in about half of these patients in the UK and abroad, and revascularisation only occurs in about half of those who have angiography. In fact, prior CABG status is an independent predictor against invasive management. Use of evidence-based drug therapies, such as aspirin, clopidogrel, ticagrelor is lower in ACS patients with prior CABG compared to in patients without prior CABG despite the fact clinical trial results suggest these drugs improve outcomes substantially in patients with prior CABG.

ISSUES AROUND THE STUDY:

PATIENT POPULATION: The study population will involve patients with an established history of coronary heart disease who have had previous CABG. Typically, CABG patients who are readmitted to hospital with recurrent angina or myocardial infarction do so at least one year after the operation (and usually 5-15 years afterwards). Therefore, these patients are usually familiar with the hospital environment and will always have had a coronary angiogram in the past since this is a requirement before CABG. Furthermore, many (e.g. at least one quarter) of these patients will have had an angioplasty in the past too. Some of these patients will have had angiograms and angioplasty procedures after the CABG also.

ISSUES RELATING TO ACUTE CORONARY SYNDROME: We will recruit patients with unstable angina or a non-ST elevation acute coronary syndrome (NSTE-ACS). These patients usually have a history of self limiting chest pain. Usually, the pain is controlled by initial medical therapy and these patients routinely wait on hospital cardiology wards often days at a time for an in-patient coronary/graft angiogram. Sometimes the angiography is deferred as an out-patient. Occasionally, angina recurs at rest or with minimal exertion (refractory ischaemia) and angiography is expedited. In the vast majority of patients, there will be ample time (minimum 4 h, usually > 24 h as appropriate) to discuss the Patient Information Sheet and obtain informed consent.

MANAGEMENT STRATEGIES: Clinical Guidelines from NICE and the European Society of Cardiology recognise that there is no evidence base to instructively inform the management of these patients thus patient and clinician preference usually inform decision-making. In this trial, patients who are invited to participate should be eligible for either treatment option. In this trial, the type of treatment in each strategy (medical or invasive) will be as per current practice in the NHS and there will be no additional study interventions. Usual care diagnostic tests including non-invasive stress testing and CT angiography may be performed if requested by the attending clinician, but these tests cannot influence the treatment group assignment of randomised patients.

HOSPITAL TYPE: A group of hospitals will be included that provide different forms of clinical services. The city hospitals in this trial will be the Western Infirmary and Glasgow Royal Infirmary. The District hospitals will be the Royal Alexandra Hospital and Royal Blackburn Hospital. One of the hospitals will have 'on-site' admission and catheterisation facilities (the Royal Blackburn Hospital) and the other hospitals participate in a regional model of care with transfer for invasive management to the regional cardiothoracic centre )the Golden Jubilee National Hospital). The standard clinical referral pathway in the NHS will be used in this trial.

OBJECTIVE OF THE PILOT: to prospectively gather information on about screening, recruitment, randomisation and initial clinical outcomes. Other than the randomisation to either medical or invasive management, the trial will essentially be observational.

RECRUITMENT: will take place during routine clinical care and will be lead by the attending clinicians who are responsible for the patients (rather than being lead by a research team).

OBJECTIVE OF THE REGISTRY: to understand the characteristics of NSTE-ACS patients with prior CABG who do not take part in the randomised trial. The reasons for not participating may be due to the presence of exclusion characteristics, patient preference, or physician preference. This information will be very important to understand feasibility and also whether or not our trial will enroll patients who are representative overall. Thus, we will record information on registry patients with prior CABG who are not randomised and follow them up in the same way as the trial patients (i.e. case note review, 1 year contact by telephone or hospital visit, electronic record linkage).

SPECIFIC AIMS RELEVANT TO DESIGN OF FUTURE DEFINITIVE CLINICAL TRIAL

PRIMARY AIMS:

1. To determine whether or not a strategy of invasive management is more effective in symptomatic patients with prior CABG compared to optimal medical therapy patients.
2. To determine whether optimal medical therapy is associated with fewer major complications and so might be safer than invasive management,
3. To prospectively quantify resource utilisation in the NHS with each treatment strategy, derive the difference in the quality-adjusted life years (QUALY) and hence evaluate comparative cost-effectiveness.

SECONDARY AIMS:

1) Quality of life (EQ-50 at baseline and 6 months); 2) components of the primary composite outcome; 3) Canadian Cardiovascular Society angina class; 4) secondary care costs.

RESEARCH HYPOTHESIS:

Unifying null hypothesis: Overall, we hypothesise that a routine invasive approach in NSTE-ACS patients with prior CABG will not be superior to a conservative non-invasive approach.

For the future multicentre definitive trial that we hope to undertake, we have adopted a pragmatic trial design. A non-inferiority trial would require a very large number of patients (and may not be ethical given the large equivalence margin), if a routine invasive approach proves not to be superior to a conservative non-invasive approach and our safety and health economic hypotheses prove correct then the trial results would support a conclusion that a routine invasive approach should not be adopted in the NHS.

Active Efficacy Hypothesis: Compared to a routine conservative non-invasive approach, an invasive approach in NSTE-ACS patients with prior CABG is associated with a lower rate of all-cause mortality, recurrent myocardial ischaemia or heart failure.

Active Safety hypothesis: Compared to an invasive approach, a conservative approach in NSTE-ACS patients with prior CABG is associated with a lower rate of adverse events related to safety during the index hospitalisation.

Health economics hypothesis: A conservative approach is associated with reduced resource utilisation compared to a routine invasive approach in NSTE-ACS patients with prior CABG.

PRIMARY AND SECONDARY ADVERSE EVENTS are defined in the Trial Protocol.

DATA MONITORING COMMITTEE - Data monitoring for safety will be coordinated by the Sponsor and Trials Unit (Pharmacovigilance).

CLINICAL EVENT COMMITTEE - A clinical event committee including 3 cardiologists independent to the research team and blind to treatment group assignment will adjudicate on the primary and secondary causes of adverse events. The case reviews will be supported with source documentation (e.g. ECGs, discharge letter, blood results), as appropriate. The adjudication decisions will be provided to the Sponsor and Clinical Trials Unit.

ELIGIBILITY:
Inclusion Criteria:

1. Unstable angina or non-ST elevation myocardial infarction
2. Stabilised symptoms without recurrent chest pain or IV therapy for 12 hrs when ambulant.

Exclusion Criteria:

1. Refractory ischaemia (i.e. recurrent angina with minimal exertion or at rest (i.e. Canadian Cardiovascular Society class III or IV) not controlled by medical therapy)
2. Cardiogenic shock
3. Inability to give informed consent
4. Unsuitable for invasive management.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
The post-randomization rate of major adverse events (co-primary composite outcome), one composite outcome for EFFICACY and one composite outcome for SAFETY. | Post randomisation, expected average followup of 1 year
  Each composite outcome (EFFICACY, SAFETY) includes major adverse events. The comparison between the incidence of each outcome according to treatment group will assess the between group difference in the proportion of major adverse events in patients allocated to non-invasive (conservative) management compared to invasive management.
  PRIMARY EFFICACY ENDPOINTS are defined as all-cause mortality, rehospitalization for refractory ischemia/angina, myocardial infarction or heart failure. The endpoints will be assessed during the study until the final randomized patient has completed 1 year follow-up. The events will be adjudicated by an independent Clinical Event Committee.
  PRIMARY SAFETY ENDPOINTS are defined as Bleeding (Bleeding Academic Research Consortium (BARC) types 2-4), stroke, procedure-related MI (Type 4a, Universal Definition), worsening renal function defined as a 25% reduction in glomerular filtration rate (GFR) or hemodialysis during the index hospitalization.

SECONDARY OUTCOMES:
Quality of life | Baseline through longer term follow-up (average follow-up 12 months
  Quality of life (Euro-quality of life 5 dimensions (EQ-5D) assessed at baseline and at 12 months
Health economics | Baseline through long term followup - average of 12 months
  Secondary care costs and procedure-related costs (diagnostic tests, PCI, CABG), hospital bed days including Intensive Care Unit, High Dependency Unit, general medical. This will be prospectively recorded for the index and any subsequent hospitalisations.
Angina severity assessment with Canadian Cardiovascular Society angina class | Baseline through long term followup - 12 months average
  Canadian Cardiovascular Society angina class will be recorded at baseline and through follow-up, average of 12 months.
Hospitalization for refractory ischemia and/or angina | Follow-up post-randomization
  Refractory Ischemia / Refractory angina are defined as recurrent ischemic symptoms lasting more than 5 minutes, while on optimal medical therapy (at least 2 anti-anginal treatments) with documented characteristic ECG changes indicative of ischaemia and requiring an additional intervention. An additional intervention was defined as reperfusion therapy for MI, cardiac catheterization, insertion of intra-aortic balloon pump or revascularization procedure (PCI or CABG surgery) within 48 hours of the onset of this episode. This definition is in line with the Timing of Intervention in Acute Coronary Syndromes (TIMACS) trial (NEJM 2009;360:2165-75).

CONTACTS AND LOCATIONS:
Overall Officials: Colin Berry, MD PhD, Principal Investigator — University of Glasgow
Locations (5):
- United Kingdom (5):
  - Royal Blackburn Hospital, Blackburn, East Lancashire
  - Royal Alexandra Hospital, Corsebar Road, Paislay, Glasgow, Scotland
  - Western Infirmary, Dumbarton Road, Glasgow
  - Glasgow Royal Infirmary, 84 Castle St, Glasgow
  - Golden Jubilee National Hospital, Clydebank, Dunbartonshire, Glasgow

REFERENCES:
- [Background] Lee MM, Petrie MC, Rocchiccioli P, Simpson J, Jackson C, Brown A, Corcoran D, Mangion K, McEntegart M, Shaukat A, Rae A, Hood S, Peat E, Findlay I, Murphy C, Cormack A, Bukov N, Balachandran K, Papworth R, Ford I, Briggs A, Berry C. Non-invasive versus invasive management in patients with prior coronary artery bypass surgery with a non-ST segment elevation acute coronary syndrome: study design of the pilot randomised controlled trial and registry (CABG-ACS). Open Heart. 2016 Apr 20;3(1):e000371. doi: 10.1136/openhrt-2015-000371. eCollection 2016. PMID 27110377
- [Background] Lee MMY, Petrie MC, Rocchiccioli P, Simpson J, Jackson CE, Corcoran DS, Mangion K, Brown A, Cialdella P, Sidik NP, McEntegart MB, Shaukat A, Rae AP, Hood SHM, Peat EE, Findlay IN, Murphy CL, Cormack AJ, Bukov NB, Balachandran KP, Oldroyd KG, Ford I, Wu O, McConnachie A, Barry SJE, Berry C; CABG-ACS Investigators. Invasive Versus Medical Management in Patients With Prior Coronary Artery Bypass Surgery With a Non-ST Segment Elevation Acute Coronary Syndrome. Circ Cardiovasc Interv. 2019 Aug;12(8):e007830. doi: 10.1161/CIRCINTERVENTIONS.119.007830. Epub 2019 Jul 31. PMID 31362541
- [Background] Lee MMY, Petrie MC, Rocchiccioli P, Simpson J, Jackson CE, Corcoran DS, Mangion K, Brown A, Cialdella P, Sidik NP, McEntegart MB, Shaukat A, Rae AP, Hood SHM, Peat EE, Findlay IN, Murphy CL, Cormack AJ, Bukov NB, Balachandran KP, Ford I, Wu O, McConnachie A, Barry SJE, Berry C; CABG-ACS Investigators. Invasive versus medically managed acute coronary syndromes with prior bypass (CABG-ACS): insights into the registry versus randomised trial populations. Open Heart. 2021 Feb;8(1):e001453. doi: 10.1136/openhrt-2020-001453. PMID 33637568
- [Background] Campbell PG, Teo KS, Worthley SG, Kearney MT, Tarique A, Natarajan A, Zaman AG. Non-invasive assessment of saphenous vein graft patency in asymptomatic patients. Br J Radiol. 2009 Apr;82(976):291-5. doi: 10.1259/bjr/19829466. PMID 19325046
- [Background] Tatoulis J, Buxton BF, Fuller JA. Patencies of 2127 arterial to coronary conduits over 15 years. Ann Thorac Surg. 2004 Jan;77(1):93-101. doi: 10.1016/s0003-4975(03)01331-6. PMID 14726042
- [Background] Sixth National Audit Cardiac Surgical Database Report (2008). Society for Cardiothoracic Surgery in Great Britain and Ireland.
- [Background] Rashid M, Ludman PF, Mamas MA. British Cardiovascular Intervention Society registry framework: a quality improvement initiative on behalf of the National Institute of Cardiovascular Outcomes Research (NICOR). Eur Heart J Qual Care Clin Outcomes. 2019 Oct 1;5(4):292-297. doi: 10.1093/ehjqcco/qcz023. PMID 31050720
- [Background] Cameron AA, Davis KB, Rogers WJ. Recurrence of angina after coronary artery bypass surgery: predictors and prognosis (CASS Registry). Coronary Artery Surgery Study. J Am Coll Cardiol. 1995 Oct;26(4):895-9. doi: 10.1016/0735-1097(95)00280-4. PMID 7560614
- [Background] Weintraub WS, Jones EL, Craver JM, Guyton RA. Frequency of repeat coronary bypass or coronary angioplasty after coronary artery bypass surgery using saphenous venous grafts. Am J Cardiol. 1994 Jan 15;73(2):103-12. doi: 10.1016/0002-9149(94)90198-8. PMID 8296729
- [Background] Mills NL, Churchhouse AM, Lee KK, Anand A, Gamble D, Shah AS, Paterson E, MacLeod M, Graham C, Walker S, Denvir MA, Fox KA, Newby DE. Implementation of a sensitive troponin I assay and risk of recurrent myocardial infarction and death in patients with suspected acute coronary syndrome. JAMA. 2011 Mar 23;305(12):1210-6. doi: 10.1001/jama.2011.338. PMID 21427373
- [Background] Elbarasi E, Goodman SG, Yan RT, Welsh RC, Kornder J, Wong GC, Dery JP, Anderson F, Gore JM, Fox KA, Yan AT; Canadian Acute Coronary Syndrome Registries I and II (ACS I and ACS II); Canadian Global Registry of Acute Coronary Events (GRACE/expanded-GRACE) Investigators. Management patterns of non-ST segment elevation acute coronary syndromes in relation to prior coronary revascularization. Am Heart J. 2010 Jan;159(1):40-6. doi: 10.1016/j.ahj.2009.09.019. PMID 20102865
- [Background] Berry C, Pieper KS, White HD, Solomon SD, Van de Werf F, Velazquez EJ, Maggioni AP, Califf RM, Pfeffer MA, McMurray JJ. Patients with prior coronary artery bypass grafting have a poor outcome after myocardial infarction: an analysis of the VALsartan in acute myocardial iNfarcTion trial (VALIANT). Eur Heart J. 2009 Jun;30(12):1450-6. doi: 10.1093/eurheartj/ehp102. Epub 2009 Apr 3. PMID 19346225
- [Background] Krumholz HM, Wang Y, Chen J, Drye EE, Spertus JA, Ross JS, Curtis JP, Nallamothu BK, Lichtman JH, Havranek EP, Masoudi FA, Radford MJ, Han LF, Rapp MT, Straube BM, Normand SL. Reduction in acute myocardial infarction mortality in the United States: risk-standardized mortality rates from 1995-2006. JAMA. 2009 Aug 19;302(7):767-73. doi: 10.1001/jama.2009.1178. PMID 19690309
- [Background] Anderson HV, Cannon CP, Stone PH, Williams DO, McCabe CH, Knatterud GL, Thompson B, Willerson JT, Braunwald E. One-year results of the Thrombolysis in Myocardial Infarction (TIMI) IIIB clinical trial. A randomized comparison of tissue-type plasminogen activator versus placebo and early invasive versus early conservative strategies in unstable angina and non-Q wave myocardial infarction. J Am Coll Cardiol. 1995 Dec;26(7):1643-50. doi: 10.1016/0735-1097(95)00404-1. PMID 7594098
- [Background] Wallentin L, Lagerqvist B, Husted S, Kontny F, Stahle E, Swahn E. Outcome at 1 year after an invasive compared with a non-invasive strategy in unstable coronary-artery disease: the FRISC II invasive randomised trial. FRISC II Investigators. Fast Revascularisation during Instability in Coronary artery disease. Lancet. 2000 Jul 1;356(9223):9-16. doi: 10.1016/s0140-6736(00)02427-2. PMID 10892758
- [Background] Cannon CP, Weintraub WS, Demopoulos LA, Vicari R, Frey MJ, Lakkis N, Neumann FJ, Robertson DH, DeLucca PT, DiBattiste PM, Gibson CM, Braunwald E; TACTICS (Treat Angina with Aggrastat and Determine Cost of Therapy with an Invasive or Conservative Strategy)--Thrombolysis in Myocardial Infarction 18 Investigators. Comparison of early invasive and conservative strategies in patients with unstable coronary syndromes treated with the glycoprotein IIb/IIIa inhibitor tirofiban. N Engl J Med. 2001 Jun 21;344(25):1879-87. doi: 10.1056/NEJM200106213442501. PMID 11419424
- [Background] Fox KA, Poole-Wilson PA, Henderson RA, Clayton TC, Chamberlain DA, Shaw TR, Wheatley DJ, Pocock SJ; Randomized Intervention Trial of unstable Angina Investigators. Interventional versus conservative treatment for patients with unstable angina or non-ST-elevation myocardial infarction: the British Heart Foundation RITA 3 randomised trial. Randomized Intervention Trial of unstable Angina. Lancet. 2002 Sep 7;360(9335):743-51. doi: 10.1016/s0140-6736(02)09894-x. PMID 12241831
- [Background] Task Force on Myocardial Revascularization of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS); European Association for Percutaneous Cardiovascular Interventions (EAPCI); Wijns W, Kolh P, Danchin N, Di Mario C, Falk V, Folliguet T, Garg S, Huber K, James S, Knuuti J, Lopez-Sendon J, Marco J, Menicanti L, Ostojic M, Piepoli MF, Pirlet C, Pomar JL, Reifart N, Ribichini FL, Schalij MJ, Sergeant P, Serruys PW, Silber S, Sousa Uva M, Taggart D. Guidelines on myocardial revascularization. Eur Heart J. 2010 Oct;31(20):2501-55. doi: 10.1093/eurheartj/ehq277. Epub 2010 Aug 29. No abstract available. PMID 20802248
- See also: Scottish Cardiac Society - Research — http://www.scottishcardiac.org/index.php?option=com_content&view=category&layout=blog&id=9&Itemid=6